CLINICAL TRIAL: NCT02784678
Title: Minimally Invasive Closed Reduction and Internal Fixation With Fully Threaded Headless Cannulated Compression Screws for Repair of Distal Radius Fracture: Study Protocol for a Randomized Controlled Trial
Brief Title: Minimally Invasive Closed Reduction and Internal Fixation With Screws for Distal Radius Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenyang Medical College (Other)
Responsible Party: Principal Investigator, Zhi Li, Director, Shenyang Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ShenyangMC_001
Record Dates: First submitted 2016-05-05; First posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures | interventions — Fracture Fixation, Internal; Open Fracture Reduction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- closed reduction group (Experimental): Patients will be assigned to C-arm fluoroscopy-assisted minimally invasive closed reduction and internal fixation with fully threaded headless cannulated compression screws (experimental group).
  Interventions: Procedure: closed reduction group
- open reduction group (Experimental): Patients will be assigned to open reduction (palmar and dorsal incisions) and internal fixation with titanium plate (control group).
  Interventions: Device: open reduction group

INTERVENTIONS:
Procedure: closed reduction group — Patients in the experimental group will undergo C-arm fluoroscopy-assisted minimally invasive closed reduction and internal fixation with fully threaded headless cannulated compression screws. In the experimental group, fractures will be reduced and internally fixed with fully threaded headless cannulated compression screws of appropriate lengths (Acutrak plus; Acumed Inc., Beaverton, OR, USA) under C-arm fluoroscopic guidance to restore the radial inclination and ulnar deviation of the distal radius.
  Other Names: minimally invasive closed reduction and internal fixation
  Arms: closed reduction group
Device: open reduction group — Patients in the control group will undergo open reduction and internal fixation with a titanium plate (Ningbo Cibei Medical Treatment Appliance Co., Ltd., Ningbo, China).
  Other Names: open reduction and internal fixation
  Arms: open reduction group

SUMMARY:
The purpose of this study is to confirm that minimally invasive closed reduction and internal fixation with fully threaded headless cannulated compression screws for distal radius fracture repair has advantages over conventional open reduction internal fixation with titanium plates, providing superior fragment stability and allowing for early rehabilitation exercise of the wrist joint, which improves recovery of function. Also to show that minimally invasive closed reduction and internal fixation with fully threaded headless cannulated compression screws is the more suitable surgical method for repair of distal radius fracture.

DETAILED DESCRIPTION:
Distal radius fracture is defined as a fracture within 3 cm of the distal articular surface. When radius fracture and ulnar styloid process fracture occur together, internal fixation is generally not pursued; however, adverse events may occur after reduction with external fixation, including unstable fracture fragments, malalignment, and loss of radial inclination and ulnar deviation, leading to wrist function impairment.

The commonly used treatment methods for distal radius fracture include internal fixation with steel plate, internal fixation with Kirschner wire, and external fixation. Open reduction and internal fixation (ORIF) has disadvantages. For example, the pronator teres is incised in palmar ORIF and in situ suturing of the muscle is not possible in most patients after implantation of the titanium plate. Even when suturing is possible, the strength of the pronator teres will decrease after surgery, and a second surgery is needed to remove the titanium plate. Dorsal ORIF is also disadvantageous because more tendons and thin soft tissue may be encountered during surgery. In addition, tendon sheath injury is inevitable, leading to myotenositis, tendon adhesion, and even tendon rupture. Thus, internal fixators should be taken out as early as possible. Satisfactory wrist function outcomes have been achieved with external fixators, in particular with dynamic external fixators. However, although external fixation has good fixing effects, it provides poor lateral stability, resulting in injury to the superficial branch of the radial nerve, screw channel infection, screw channel fracture, screw loosening, and even Sudeck's atrophy. Internal fixation with Kirschner wire generates minimal surgical trauma, but this technique does not provide sufficient strength for fixation and is therefore rarely used at present. There is an urgent need to develop a more stable fixation method for distal radius fracture. Minimally invasive surgery avoids the tissue damage and impairment of physiological function caused by open surgery because of its precise location techniques. Brachial plexus anesthesia allows surgeons to avoid large incisions and excessive bleeding. There are no palmar or dorsal incisions in minimally invasive surgery for distal radius fractures, so the structures surrounding the wrist joint are not iatrogenically damaged, which theoretically improves wrist function recovery.

During C-arm fluoroscopy-assisted minimally invasive closed reduction, either no surgical incision or an incision only 0.5 cm in length is made at the wrist joint; the fracture fragments are reduced with fully threaded headless cannulated compression screws. Repair stability is assessed with the C-arm fluoroscopic X-ray system. This method is theoretically feasible for distal radius fractures. The fracture fragments are fixed with fully threaded, cannulated, variable-pitch, headless compression screws, which can increase fragment stability. Therefore, the investigators hypothesize that C-arm fluoroscopy-assisted minimally invasive closed reduction will fix distal radius fractures and allow patients to perform wrist function exercises as early as possible.

Our previous studies have confirmed that minimally invasive closed reduction and internal fixation with fully threaded headless cannulated compression screws has precise therapeutic effects for distal radius fractures. This method can improve wrist function, and has therapeutic effects similar to those of conventional open reduction and internal fixation with titanium plates. The results of these previous studies are shown in Table 1. However, it is not clear whether minimally invasive closed reduction and internal fixation with fully threaded headless cannulated compression screws has advantages over conventional open reduction and internal fixation with titanium plates for distal radius fracture repair.

In this study, the investigators hypothesized that minimally invasive closed reduction and internal fixation with fully threaded headless cannulated compression screws provides better stability than conventional methods, and can effectively promote the early recovery of wrist function. Under conditions of no cutting of fracture fragments, no blood supply compromise in the fracture fragments, and no destruction of the local microenvironment, and with C-arm fluoroscopy assistance, the investigators will perform minimally invasive closed reduction, pressurizing the fracture fragments with fully threaded headless cannulated compression screws, and will investigate whether this method of distal radius fracture repair provides satisfactory stability and allows early wrist function recovery.

Safety assessment Adverse events should be accurately recorded, including time of onset, severity, duration, and measures taken. The known possible adverse events include bone nonunion, displaced fracture, wrist joint pain, Sudeck's syndrome, primary or secondary tendon injury, shoulder-hand syndrome, traumatic arthritis of the wrist joint, implant failure, malunion, infection, septicemia, and thrombosis.

Any of the following will be considered a severe adverse event: death, prolonged hospital stay, mutilation, fatal reaction, or teratogenicity. Any adverse event occurring during the trial will be reported to the researchers in charge and to the ethics committee within 24 hours.

Data management Data from the trial will be kept in a secure, locked storage area with limited access for later review by a biostatistician, a researcher in charge.

Statistical analysis All data will be statistically processed with SPSS 11.0 software (SPSS, Chicago, IL, USA). Normally distributed measurement data will be expressed as mean and SD. Non-normally distributed measurement data will be expressed as lower quartile (q1), median, and upper quartile (q3). The numeration data will be expressed as constituent ratios. The Mann-Whitney U non-parametric test will be used to compare age and course of disease between the experimental and control groups. The chi-square test will be used to compare sex differences between the two groups. The Mann-Whitney U non-parametric test will also be used to compare imaging parameters (for example, angle, height, and length), PRWE scores, healing time of fracture, and VAS scores. The chi-square test will also be used to compare the effective rate between the two groups. An alpha level of 0.05 (two-sided) will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years or older, either sex
* A history of known trauma
* Presence of wrist joint pain and limitation of motion after trauma
* Fracture occurring 2.0-3.0 cm proximal to the articular surface, confirmed with imaging findings
* Unstable distal radius fracture
* Dorsal displacement of fracture fragment
* Fracture involving the wrist joint, but no more than two fracture fragments involving the wrist joint

Exclusion Criteria:

* Acute fracture of several other regions, including the ulnar styloid process
* Open fracture
* Mental disorder
* Occurrence of fracture more than 21 days before presentation
* Severe heart, lung, liver, or kidney function disorder
* Severe local infection after fracture
* Refusal to sign informed consent form
* Poor compliance, or upon the request of the sponsor for safety reasons
* If participation in the trial would be a potential hazard to patient's health

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
change of X-ray findings | Baseline and week 3, week 6, week 12, week 24 after surgery
  X-ray findings to evaluate fracture healing

SECONDARY OUTCOMES:
change of CT findings | Baseline and week 3, week 6, week 12, week 24 after surgery
  CT findings to evaluate fracture healing
change of patient-rated wrist evaluation score results | week 3, week 6, week 12, week 24 after surgery
  Patient-rated wrist evaluation score to evaluate wrist joint function
change of healing of fracture | week 3, week 6, week 12, week 24 after surgery
  earlier radiographic disappearance of the fracture line indicates faster healing
change of Visual Analogue Scale(VAS) score | week 3, week 6, week 12, week 24 after surgery
  Visual Analogue Scale(VAS) score is used to evaluate wrist joint pain after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Li, Master, Principal Investigator — Department of Orthopedic Surgery, Central Hospital Affiliated to Shenyang Medical College, Shenyang, Liaoning Province, China

IPD SHARING:
Plan to Share IPD: Undecided